CLINICAL TRIAL: NCT06795061
Title: A Fitness Buddy Program to Boost University Students' Physical Activity Levels
Brief Title: Fitness Buddy Program to Boost Physical Activity in University Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinan University Guangzhou (Other)
Responsible Party: Principal Investigator, Ma Ruisi, lecturer, Jinan University Guangzhou
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBRE-24-0228; TDLEG (Other Grant/Funding Number: the Chinese University of Hong Kong)
Record Dates: First submitted 2025-01-24; First posted 2025-01-27 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Physical Inactivity; Psychological Stress; Mental Well-being
MeSH Terms: conditions — Sedentary Behavior; Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer-Supported Exercise Group (Experimental): Participants will form peer-support groups of four to six students. They will coordinate weekly exercise sessions (e.g., running, cycling, yoga), share goals, and encourage each other. A professional coach provides knowledge-based guidance on exercise safety, basic nutrition, and motivation strategies, but does not conduct in-person training.
  Interventions: Behavioral: Peer-Supported Exercise with Professional Guidance
- Control Group (Usual Campus Resources) (No Intervention): Participants will have access to the usual resources available on campus (e.g., sports facilities, counseling services) without any structured peer-support exercise sessions or professional coaching.

INTERVENTIONS:
Behavioral: Peer-Supported Exercise with Professional Guidance — Participants will engage in small, peer-supported exercise groups (4-6 individuals) to coordinate weekly sessions (e.g., running, cycling, yoga). A professional coach provides knowledge-based guidance remotely, focusing on safe exercise techniques, injury prevention, basic nutrition, and motivation strategies, but does not conduct in-person training sessions. The aim is to improve adherence to physical activity and enhance mental well-being through peer accountability and evidence-informed coaching.
  Arms: Peer-Supported Exercise Group

SUMMARY:
This study explores whether a peer-supported "fitness buddy" program can help first-year university students increase physical activity levels and improve mental well-being. Over 12 weeks, participants will form small exercise groups, choose enjoyable activities (such as jogging, cycling, or yoga), and support each other through shared goals and regular check-ins. A professional coach will offer weekly guidance on exercise safety, injury prevention, and motivation strategies, but the actual workouts will be conducted by the students.

The investigators aim to determine if this peer-based approach helps reduce stress, anxiety, and depressive symptoms, while boosting self-esteem and social connectedness. Students in a control group will receive usual campus resources without structured group support. By comparing outcomes at the start, after the 12-week program, and again at follow-up, the study will assess whether peer-led, knowledge-supported exercise can sustainably enhance both physical and mental health during the critical transition into university life.

DETAILED DESCRIPTION:
This longitudinal, parallel-group study focuses on first-year undergraduates (ages 18-25) who are not currently engaged in structured exercise programs. Participants meeting inclusion criteria will be assigned to either a peer-supported exercise group (with weekly professional guidance) or a control group (usual campus resources, no structured group sessions). The peer-support model encourages accountability, shared goal-setting, and regular communication via group messaging tools.

Data collection will include physical activity levels (e.g., International Physical Activity Questionnaire), mental health outcomes (GAD-7, PHQ-9), perceived stress (PSS), self-esteem (RSES), loneliness (UCLA Loneliness Scale), and social connectedness (SCS). Assessments occur at baseline, 12 weeks (post-intervention), and at a short-term follow-up (Week 16) to evaluate both immediate and sustained effects. All participants will receive instructions on safe exercise practices. Potential risks, such as minor injuries or discomfort discussing mental health, will be minimized through clear guidance, optional campus support resources, and respect for privacy. The findings may help universities develop targeted programs that combine knowledge-based coaching with peer support to enhance students' physical and psychosocial well-being.

ELIGIBILITY:
Inclusion Criteria

1. First-year undergraduate students (ages 18-25) enrolled at the university.
2. Able to safely participate in moderate-intensity exercise as determined by a pre-screening health questionnaire.
3. Willing to join a 12-week, peer-supported exercise program and complete all baseline, post-intervention, and follow-up assessments.

Exclusion Criteria

1. Documented medical conditions that preclude safe engagement in moderate-intensity physical activity (e.g., severe cardiovascular disease, uncontrolled hypertension).
2. Current major psychiatric disorders (e.g., psychotic disorders) that could significantly impede adherence to the study protocol.
3. Enrollment in any structured exercise program (≥3 sessions per week) for at least 3 consecutive months prior to study entry.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Activity Levels (IPAQ) | Baseline, Week 12 (post-intervention), and Week 16 (follow-up)
  Self-reported physical activity levels will be assessed using the International Physical Activity Questionnaire (IPAQ), capturing frequency, duration, and intensity of exercise. This will help determine whether peer-supported exercise plus professional guidance leads to significant changes in overall activity compared to usual campus resources.

SECONDARY OUTCOMES:
Change in Overall Mental Health and Psychosocial Well-Being | Baseline, Week 12 (post-intervention), and Week 16 (follow-up)
  Mental health and psychosocial well-being will be evaluated using multiple standardized questionnaires, including the Generalized Anxiety Disorder Scale (GAD-7), the Patient Health Questionnaire (PHQ-9) for depressive symptoms, the Perceived Stress Scale (PSS), the Rosenberg Self-Esteem Scale (RSES), the UCLA Loneliness Scale, and the Social Connectedness Scale (SCS). Composite changes across these measures will be used to assess overall psychosocial functioning over the course of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Education Unit, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including demographic information and outcome measures) will be made available to qualified researchers upon reasonable request. A data use agreement (DUA) must be signed, and approval from our institutional ethics committee may be required. Data will be made available after publication of the primary findings and for up to 5 years thereafter.